CLINICAL TRIAL: NCT04624035
Title: Comparison Between Implantable Phakic Intraocular Lens and Implantable Collamer Lens in Treatment of Myopia in Adults
Brief Title: Implantable Phakic Lens (IPCL) VS Implantable Collamer Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud F. Rateb, Associate professor of ophthalmology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICL vs IPCL
Record Dates: First submitted 2020-10-20; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantable Collamer Lens (ICL, V4c with central hole) in treatment of myopia in adults. (Active Comparator): Implantation of ICL (V4c with central hole) for treatment of myopia in adults using peribulbar anesthesia. Thirty minutes before surgery, cycloplegic and phenylephrine eye drops were applied. Five minutes before surgery, povidone-iodine 5% was applied. The anterior chamber was filled with sodium hyaluronate 1%, which was completely removed at the end of the surgery. The lens was inserted using the ICL injector. Tobramycin and dexamethasone 0.1% eye drops were used four times a day for 10 days, after which diclofenac sodium eye drops were started four times a day for 2 weeks.
  Interventions: Procedure: Implantable Collamer Lens (ICL) in treatment of myopia in adults.
- Acrylic Implantable Intraocular Lens (IPCL, V2) in treatment of myopia in adults (Active Comparator): Implantation of IPCL for treatment of Myopia in adults using peribulbar anesthesia. Thirty minutes before surgery, cycloplegic and phenylephrine eye drops were applied. Five minutes before surgery, povidone-iodine 5% was applied. The anterior chamber was filled with sodium hyaluronate 1%, which was completely removed at the end of the surgery. The lens was inserted using the IPCL injector. Tobramycin and dexamethasone 0.1% eye drops were used four times a day for 10 days, after which diclofenac sodium eye drops were started four times a day for 2 weeks.
  Interventions: Procedure: Implantable Intraocular Lens (IPCL) in treatment of myopia in adults.

INTERVENTIONS:
Procedure: Implantable Collamer Lens (ICL) in treatment of myopia in adults. — ICL Group: After mydriatic eye drops and topical anesthesia instillation, a 3-mm temporal corneal incision was done. Viscoelastic material was injected in the anterior chamber (AC). An injector cartridge (STAAR Surgical) was used to insert the ICL V4c model with central hole). The four footplates of the ICL were positioned on the ciliary sulcus at the 180° axis. Viscoelastic material was entirely taken away.
  Other Names: All drugs used were mentioned in the arm description
  Arms: Implantable Collamer Lens (ICL, V4c with central hole) in treatment of myopia in adults.
Procedure: Implantable Intraocular Lens (IPCL) in treatment of myopia in adults. — IPCL Group: Topical anesthetic and mydriatic agents were instilled before surgery. Using peripulbar anaesthesia, the IPCL (V2 model with central hole) was implanted into the AC through a 3 mm clear corneal incision after viscoelastic material injection. The footplates were subsequently tucked behind the iris, followed by a thorough viscoelastic removal.
  Other Names: All drugs used were mentioned in the arm description
  Arms: Acrylic Implantable Intraocular Lens (IPCL, V2) in treatment of myopia in adults

SUMMARY:
Phakic intraocular lenses (pIOL) of different designs and materials have been used effectively instead of corneal refractive surgery in certain situations. The pIOL exhibits a number of advantages over corneal techniques as it is suitable for high myopes, with lower production of aberrations, and superior contrast sensitivity. Keeping the accommodation is its definite lead over refractive lens exchange. The Visian implantable collamer lens (ICL; Staar Surgical, Monrovia, CA), a posterior chamber pIOL, has been stated to be useful for the correction of high myopia. Nevertheless, as an intraocular procedure, it is associated with a risk of complications as probable injury to anterior segment, retinal detachment and endophthalmitis.

The Implantable Phakic Contact Lens (IPCL V2, Caregroup Sight Solutions, India) has been developed as an alternative for the ICL, at a noticeable financial advantage. Furthermore, the highestmyopic correction which is instantly accessible with ICL is -18.0 D. Meanwhile, IPCL can provide correction higher degrees up to -30.0 D.

Former researches have been made to assess the safety and efficiency of ICL implantation, to evaluate various devices for anterior segment imaging postoperatively and to identify changes in anterior segment after surgery. A recent study determined the safety of the IPCL over a minimum follow-up period of one year. In this work the investigators aimed to compare the refractive results and the adverse effects of the IPCL and the ICL in treatment of myopia in adults.

ELIGIBILITY:
Inclusion Criteria:

* myopia of more than 6 diopter
* central anterior chamber depth more than 2.8 mm

Exclusion Criteria:

* unstable refraction
* any other ocular disease
* any systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Refractive outcome | 12 months
  Postoperative refractive error measured in spherical equivalent
Visual outcome | 12 months
  Uncorrected distance and near vision using Snellen's chart and using decimal fractions

SECONDARY OUTCOMES:
Adverse reactions | 12 months
  adverse reactions will be recorded including intraocular inflammation, corneal endothelial changes and lens opactification

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud F Rateb, MD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Tiba eye center, Asyut
  - Al Masa eye center, Banhā

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underline the results of this trial will be available once completion of the study after de-identification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 month and ending 36 months after trial publication
Access Criteria: for individual participant data meta-analysis

REFERENCES:
- [Background] Stulting RD, John ME, Maloney RK, Assil KK, Arrowsmith PN, Thompson VM; U.S. Verisyse Study Group. Three-year results of Artisan/Verisyse phakic intraocular lens implantation. Results of the United States Food And Drug Administration clinical trial. Ophthalmology. 2008 Mar;115(3):464-472.e1. doi: 10.1016/j.ophtha.2007.08.039. Epub 2007 Nov 26. PMID 18031820
- [Background] Kamiya K, Igarashi A, Shimizu K, Matsumura K, Komatsu M. Visual performance after posterior chamber phakic intraocular lens implantation and wavefront-guided laser in situ keratomileusis for low to moderate myopia. Am J Ophthalmol. 2012 Jun;153(6):1178-86.e1. doi: 10.1016/j.ajo.2011.12.005. Epub 2012 Feb 23. PMID 22365084
- [Background] Sanders D, Vukich JA. Comparison of implantable collamer lens (ICL) and laser-assisted in situ keratomileusis (LASIK) for low myopia. Cornea. 2006 Dec;25(10):1139-46. doi: 10.1097/ICO.0b013e31802cbf3c. PMID 17172886
- [Background] Igarashi A, Kamiya K, Shimizu K, Komatsu M. Visual performance after implantable collamer lens implantation and wavefront-guided laser in situ keratomileusis for high myopia. Am J Ophthalmol. 2009 Jul;148(1):164-70.e1. doi: 10.1016/j.ajo.2009.02.001. Epub 2009 Apr 17. PMID 19375059
- [Background] Pineda-Fernandez A, Jaramillo J, Vargas J, Jaramillo M, Jaramillo J, Galindez A. Phakic posterior chamber intraocular lens for high myopia. J Cataract Refract Surg. 2004 Nov;30(11):2277-83. doi: 10.1016/j.jcrs.2004.03.035. PMID 15519075
- [Background] Elmohamady MN, Abdelghaffar W. Anterior Chamber Changes After Implantable Collamer Lens Implantation in High Myopia Using Pentacam: A Prospective Study. Ophthalmol Ther. 2017 Dec;6(2):343-349. doi: 10.1007/s40123-017-0109-3. Epub 2017 Sep 20. PMID 28933042
- [Background] Fernandes P, Gonzalez-Meijome JM, Madrid-Costa D, Ferrer-Blasco T, Jorge J, Montes-Mico R. Implantable collamer posterior chamber intraocular lenses: a review of potential complications. J Refract Surg. 2011 Oct;27(10):765-76. doi: 10.3928/1081597X-20110617-01. Epub 2011 Jun 30. PMID 21710954
- [Background] Sachdev G, Ramamurthy D. Long-term safety of posterior chamber implantable phakic contact lens for the correction of myopia. Clin Ophthalmol. 2019 Jan 7;13:137-142. doi: 10.2147/OPTH.S185304. eCollection 2019. PMID 30662257
- [Background] Zhang J, Luo HH, Zhuang J, Yu KM. Comparison of anterior section parameters using anterior segment optical coherence tomography and ultrasound biomicroscopy in myopic patients after ICL implantation. Int J Ophthalmol. 2016 Jan 18;9(1):58-62. doi: 10.18240/ijo.2016.01.10. eCollection 2016. PMID 26949611
- [Derived] Rateb M, Gad AAM, Tohamy D, Elmohamady MN. A Prospective Comparative Study between Implantable Phakic Intraocular Contact Lens and Implantable Collamer Lens in Treatment of Myopia in Adults. J Ophthalmol. 2022 Mar 28;2022:9212253. doi: 10.1155/2022/9212253. eCollection 2022. PMID 35388352